CLINICAL TRIAL: NCT05326373
Title: A Pilot Study to Evaluate Gingivitis Using Traditional and Molecular Methods
Brief Title: Stannous Fluoride and Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022001
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Tin Fluorides

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Group (Active Comparator): Subjects without gingivitis (</= 3 bleeding sites) will use stannous fluoride toothpaste
  Interventions: Drug: Stannous fluoride
- Unhealthy Group (Active Comparator): Subjects with gingivitis (>/= bleeding 20 sites) will use stannous fluoride toothpaste
  Interventions: Drug: Stannous fluoride

INTERVENTIONS:
Drug: Stannous fluoride — brush twice daily with stannous fluoride toothpaste for 8 weeks

SUMMARY:
8-week study using stannous fluoride toothpaste on subjects with gingivitis ("unhealthy") and without gingivitis ("healthy"). Gingivitis index will be performed at BL, Week 4 and Week 8. A number of biological samples will be collected at each timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older;
* Provide written informed consent and receive a signed copy of consent;
* Agree to delay any elective dentistry, including dental prophylaxis, and to report any non-study dentistry received during the course of this study;
* Agree not to participate in any other oral care studies for the duration of this study;
* Agree to refrain from any form of non-specified oral hygiene during the treatment periods, including but not limited to the use of products such as floss or whitening products;
* Agree to return for all scheduled visits and follow study procedures;
* Have at least 16 natural teeth;
* Be in good general health, as determined by the Investigator/designee based on a review of the health history/update for participation in the study.

For Unhealthy Group:

* Have at least 20 bleeding sites (sites with a score of 1 or 2 on the Screening GBI exam); and
* Have a minimum of 3 sampling sites with bleeding and pocket depth >/=3mm but not deeper than 4mm at the Screening visit.

For Healthy Group:

* Have a maximum of 3 bleeding sites (sites with a score of 1 or 2 on the Screening GBI exam); and
* No pockets deeper than 2mm.

Exclusion Criteria:

* Self-reported pregnancy or the intent to become pregnant anytime during the course of the study;
* Inability to comply with study procedures;
* Rampant caries, open or untreated caries, or advanced periodontitis requiring prompt treatment;
* Severe periodontal disease, including but not limited to purulent exudate, generalized mobility, and/or severe recession;
* Fixed orthodontic appliances or attachments for aligner treatment;
* Having had a dental prophylaxis within 2 weeks of plaque sampling visits;
* Having taken antibiotics or used anti-gingivitis/anti-bacterial oral care products such as chlorhexidine or Listerine within 2 weeks of plaque sampling visits;
* Needing an antibiotic prophylaxis prior to dental visits;
* Presenting with any disease or condition(s) that could be expected to interfere with examination procedures or the subject's safe completion of the study; or
* Having any condition or disease, as determined by the Investigator/Designee which could be expected to interfere with examination procedures or with the subject's safe completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
MGI | 8 weeks
  Modified Gingival Index- validated assessment of gingival health looking at inflammation based on 4-point range 0 (normal gingiva) to 4 (severe inflammation).
GBI | 8 weeks
  Gingival Bleeding Index- validated assessment of gingival health looking at bleeding based on 2-point range 0 (Absence of bleeding) to 2 (Immediate bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

REFERENCES:
- [Derived] Ramji N, Xie S, Bunger A, Trenner R, Ye H, Farmer T, Reichling T, Ashe J, Milleman K, Milleman J, Klukowska M. Effects of stannous fluoride dentifrice on gingival health and oxidative stress markers: a prospective clinical trial. BMC Oral Health. 2024 Aug 30;24(1):1019. doi: 10.1186/s12903-024-04785-7. PMID 39215289